CLINICAL TRIAL: NCT00737399
Title: Anxiety and Depression Levels in Cancer Patients After Self-Application of EFT (Emotional Freedom Techniques)
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Soul Medicine Institute (Other)
Responsible Party: Principal Investigator, Dawson Church, Principal Investigator, Soul Medicine Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SMI-CHOL-82008
Record Dates: First submitted 2008-08-18; First posted 2008-08-19 (Estimated); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Depression
Keywords: depression; anxiety; pain; insomnia; cancer; cholangiocarcinoma; EFT (Emotional Freedom Techniques)
MeSH Terms: conditions — Depression; Anxiety Disorders; Pain; Sleep Initiation and Maintenance Disorders; Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Lifestyle Counseling with Emotional Freedom Techniques (EFT)
  Interventions: Behavioral: Lifestyle Counseling with Emotional Freedom Techniques (EFT)

INTERVENTIONS:
Behavioral: Lifestyle Counseling with Emotional Freedom Techniques (EFT) — Two series of four sessions of phone support group coaching instruction in the use of EFT

SUMMARY:
Anxiety and depression have been found to be significant co-occurring conditions in cancer patients. This study examines these and other psychological conditions in patients diagnosed with cholangiocarcinoma, a rare cancer of the bile duct, with an average survival time of three to six months post-diagnosis. Participants are taught EFT in telephone and internet group coaching sessions, and have access to an online support forum. They complete the Mini-Mental Adjustment to Cancer Scale (Mini-MAC), EORTC Quality of Life scale, the PTSD checklist, the Patient Health Questionnaire, and a brief health checklist. Participants also provide medical records confirming their diagnosis, and markers, both before and after the study. The study is expected to enroll 20-15 cholangiocarcinoma patients, and use a within-subjects, time series, repeated measures design. Symptoms are assessed prior to coaching, after four, and again after eight weekly coaching sessions. Follow-ups will occur in one month, three months, and one year. It is hypothesized that a drop in the severity of co-occurring psychological symptoms, pain and insomnia may occur after EFT coaching.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cholangiocarcinoma
* Ability to complete forms and attend phone coaching sessions

Exclusion Criteria:

* None

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2008-09; Primary Completion 2028-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
depression | duration of study

SECONDARY OUTCOMES:
anxiety | duration of study
pain | duration of study
insomnia | duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Dawson Church, PhD, Principal Investigator — Soul Medicine Institute
Locations (1):
- Soul Medicine Institute, Santa Rosa, California, United States

REFERENCES:
- [Background] Endo I, Gonen M, Yopp AC, Dalal KM, Zhou Q, Klimstra D, D'Angelica M, DeMatteo RP, Fong Y, Schwartz L, Kemeny N, O'Reilly E, Abou-Alfa GK, Shimada H, Blumgart LH, Jarnagin WR. Intrahepatic cholangiocarcinoma: rising frequency, improved survival, and determinants of outcome after resection. Ann Surg. 2008 Jul;248(1):84-96. doi: 10.1097/SLA.0b013e318176c4d3. PMID 18580211
- See also: Cholangiocarcinoma Foundation — http://cholangiocarcinoma.org